CLINICAL TRIAL: NCT05279300
Title: A Phase I, Dose-Escalation and Dose-Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activities of CS5001, an Anti-ROR1 Antibody-Drug Conjugate, Used as A Single Agent and in Combination With Systemic Therapies in Patients With Advanced Solid Tumors and Lymphomas
Brief Title: A Study of CS5001 in Patients With Advanced Solid Tumors and Lymphomas
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: CStone Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CS5001-101
Record Dates: First submitted 2022-03-04; First posted 2022-03-15 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor; Advanced Lymphoma
MeSH Terms: interventions — Rituximab; Gemcitabine; Oxaliplatin; Lenalidomide; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dose escalation (Experimental)
  Interventions: Drug: CS5001
- Dose expansion (Experimental)
  Interventions: Drug: CS5001; Biological: Rituximab; Drug: Gemcitabine; Drug: Oxaliplatin; Drug: Lenalidomide; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Prednisone

INTERVENTIONS:
Drug: CS5001 — The dose and dosing schedule is decided by the Safety Monitoring Committee.
Biological: Rituximab — IV infusion
  Arms: Dose expansion
Drug: Gemcitabine — IV infusion
  Arms: Dose expansion
Drug: Oxaliplatin — IV infusion
  Arms: Dose expansion
Drug: Lenalidomide — PO
  Arms: Dose expansion
Drug: Cyclophosphamide — IV infusion
  Arms: Dose expansion
Drug: Doxorubicin — IV infusion
  Arms: Dose expansion
Drug: Vincristine — IV infusion
  Arms: Dose expansion
Drug: Prednisone — PO
  Arms: Dose expansion

SUMMARY:
This is a first-in-human (FIH) study to evaluate the safety and preliminary efficacy of experimental drug CS5001 used as a single agent and in combination with systemic therapies in patients with advanced hematological and solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* For solid tumor patients of dose escalation, they must have pathologically confirmed, unresectable advanced solid tumor with disease progression on or after at least 1 line of prior systemic therapy.
* For Lymphoma patients of dose escalation, they must have pathologically confirmed Hodgkin and non-Hodgkin B-cell lymphoma as defined per 2016 World Health Organization(WHO) classification, with disease progression on or after at least 2 lines of prior systemic therapy.
* For mono-therapy cohorts, eligible patients must have pathologically confirmed relapsed/refractory (R/R) lymphomas or advanced solid tumors, and have demonstrated failure with previous line(s) of standard-of-care treatment. Patients in the solid tumor cohort must exhibit ROR1-positive expression in their baseline tumor tissues. For combination therapy cohorts, DLBCL patients must either be treatment-naïve or have experienced failure with at least one prior line of standard-of-care therapy to qualify for treatment with CS5001 in combination with first-line or subsequent standard-of-care therapies for DLBCL. Solid tumor patients must have pathologically confirmed disease, be naïve to PD-1/PD-L1 inhibitors, and have at least failed first-line therapy or standard-of-care treatment.
* For dose escalation, with at least one evaluable lesion as defined per Response Evaluation Criteria in Solid Tumours(RECIST) v1.1 solid tumor or per 2014 Lugano Classification Criteria for lymphoma, respectively. For dose expansion, with at least one measurable lesion as defined per RECIST v1.1 solid tumor or per 2014 Lugano Classification Criteria for lymphoma, respectively.
* Life expectancy > 3 months.
* Eastern Cooperative Oncology Group(ECOG) performance status 0-2.
* Have adequate organ function.

Exclusion Criteria:

* Has disease that is suitable for local treatment administered with curative intent. For lymphoma, candidacy for hematopoietic stem cell transplantation based on the Investigator's judgment.
* Has a history of a second malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured.
* For dose expansion: Participation in other studies involving therapies targeting ROR1 prior to study entry and/or during study participation.
* Has known central nervous system (CNS) lymphoma or solid tumor CNS metastasis that is either symptomatic, untreated, or requires therapy.
* Has other acute or chronic medical or psychiatric conditions.
* Has a diagnosis of immunodeficiency, or has an active autoimmune disease or other conditions that require systemic steroid therapy.
* Has peripheral edema, pericardial effusion, or ascites indicated for medical intervention or limiting activity of daily life. Or with a known history of peripheral vasculopathies.
* Patients with any active infections requiring systemic therapy within 2 weeks prior to the administration of the first dose of the study drug.
* Patients known to be human immunodeficiency virus (HIV)-positive or have acquired immune deficiency syndrome (AIDS).
* Significant cardiovascular disease within 6 months prior to the first dose of the study drug.
* Significant screening electrocardiogram (ECG) abnormalities.
* Has received major surgery, chemotherapy, definitive radiotherapy, target therapy, immunotherapy, or other anti-cancer therapy within 21 days prior to the administration of the first dose of the study drug.
* Administration of a live vaccine within 28 days prior to the administration of the first dose of the study drug.
* Has active graft versus host disease.
* With known active alcohol or drug abuse.
* Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of CS5001 if any (for dose escalation part) | About 6 months
  Participants will receive CS5001 for injection once every three weeks. The MTD will be determined by the number of participants who experience a dose limiting toxicity (DLT).
Recommended Phase 2 Dose(RP2D) of CS5001 (for dose escalation part) | About 6 months
  The selection of RP2D will be based on consideration of overall safety information together with available pharmacokinetic, pharmacodynamic, and efficacy data. The RP2D may be the MTD or may be a lower dose within the tolerable dose range.
Incident and severity of adverse events | Until 90 days since the last dose of investigational product or until initiation of a new anti-cancer treatment, whichever occurs first
Objective Response Rate (ORR) (for dose expansion) | Up to 2 years
  The percentage of participants with a CR or PR based on 2014 Lugano Classification Criteria for lymphomas, iwCLL 2018 guidelines for CLL/SLL and RECIST v1.1 for solid tumors.

SECONDARY OUTCOMES:
Concentration of CS5001 total antibody | Up to 30 days since the last dose of or until initiation of a new anti-cancer treatment, whichever occurs first
Concentration of anti-CS5001 antibodies | Up to 30 days since the last dose of or until initiation of a new anti-cancer treatment, whichever occurs first

OTHER OUTCOMES:
Anti-tumor activity of CS5001 at RP2D in patient with selected advanced cancers (For dose expansion part) | About up to 12 months

CONTACTS AND LOCATIONS:
Locations (37):
- United States (3):
  - North Shore Hematology Oncology Associates, East Setauket, New York
  - Columbia U. - Herbert Irving Comprehensive Cancer Center, New York, New York
  - BUMC - Mary Crowley Cancer Research Centers (MCCRC), Dallas, Texas
- Australia (6):
  - Scientia Clinical Research Limited, Randwick, New South Wales
  - Ashford Cancer Centre Research, Adelaide, South Australia
  - Central Adelaide Local Health Network Incorporated, Adelaide, South Australia
  - Royal Adelaide Hospital (RAH), Adelaide, South Australia
  - Epworth Freemasons Medical Centre, East Melbourne, Victoria
  - Epworth Foundation trading as Epworth HealthCare, Melbourne, Victoria
- China (28):
  - Anhui Provincial Cancer Hospital, Hefei, Anhui
  - Anhui Provincial Hospital,, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Yanda Lu Dao Pei Hospital, Beijing, Beijing Municipality
  - The Cancer Hospital Affiliated to Chongqing University, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Guangdong Province Hospital, Guangzhou, Guangdong
  - Sun YatSen University Cancer Center, Guangzhou, Guangdong
  - Guangxi Medical University Affiliated Tumour Hospital, Nanning, Guangxi
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu province hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhu, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - The first Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Fudan University Shanghai Cancer Hospital, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No